CLINICAL TRIAL: NCT03339700
Title: Addition of Gemcitabine to the Standard Reduced Busulfan and Cyclophosphamide (BUCY2) Pre Allogeneic Hematopoietic Stem Cell Transplantation Conditioning for Acute Lymphoblastic Leukemia
Brief Title: Addition of Gemcitabine to Pre Allo-HSCT Conditioning for Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMNSZ REF 2235
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Gemcitabine; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unique (Experimental): Patients will receive reduced Busulfan and Cyclophosphamide (BUCY 2) conditioning regimen, consisting in the administration of two medications: Busulfan and Cyclophosphamide Plus: Gemcitabine. Then patients will undergo an Allogeneic Hematopoietic Stem Cell Transplantation.
  Interventions: Drug: Gemcitabine; Drug: Busulfan; Drug: Cyclophosphamide; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Gemcitabine — 4800mg/m2, intravenous (IV), divided 4 days, 1200mg/m2/day, during days -5 to -2
  Other Names: Gemzar
Drug: Busulfan — 12mg/kg, Oral, divided in 4 days, 3mg/kg/day Oral, during days -7 to -4.
  Other Names: Myleran
Drug: Cyclophosphamide — 80mg/kg, intravenous (IV), divided in 2 days, 40mg/kg/day IV, during days -3 and -2.
  Other Names: Cytoxan
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Bone Marrow HSC (allogeneic HSCT) transfusion, day 0
  Other Names: Allogeneic Bone Marrow Transplantation

SUMMARY:
The main purpose of the project is to evaluate the disease free survival and overall survival in patients diagnosed with acute lymphoblastic leukemia undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT) adding gemcitabine to the standard institutional conditioning regimen based on two alkylating drugs, reduced busulfan and cyclophosphamide (reduced BUCY 2).

DETAILED DESCRIPTION:
In the last decade, hematopoietic stem cell transplantation (HSCT) has become an efficient strategy for the treatment of high risk acute lymphoblastic leukemias. Lymphoid acute leukemias (ALL) are considered malignant clonal diseases of the hematopoietic stem cells, and represent a therapeutic challenge due to the high relapse rate and mortality using conventional chemotherapy regimens. Many studies have shown a decrease in relapse and an increase in overall survival with allogeneic HSCT, however, despite the fact that results in ALL have improved in the past years, achieving complete remission (CR) in approximately 75% of the patients, the relapse rate remains high and long term survival is lower than 50% depending on age and disease characteristics. On the other hand, it has been stated that relapse is higher when an allo-HSCT is performed in second CR, obtaining poorer results compared to performing HSCT in first CR, although better than chemotherapy alone (87% probability of relapse).

It is necessary to implement strategies that increase efficiency of pre transplant conditioning regimens in patients diagnosed with ALL undergoing an allo-HSCT in order to reduce relapse and increase overall survival. The hypothesis is that adding gemcitabine to the standard institutional conditioning regimen (reduced BUCY 2) in patients with ALL undergoing an allo-HSCT, the relapse free survival as well as the overall survival will improve, because it has been demonstrated in other malignant hematological diseases that gemcitabine plus two alkylating agents, facilitates synergism with busulfan and melphalan, inhibiting the DNA damage repair and causing a higher cytotoxic effect.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia in 2nd complete remission or primary refractory disease, candidates to hematopoietic stem cell transplantation.
* Hemoglobin ≥ 10 g/dl, Absolute Neutrophil Count ≥ 1 x 103/mm3, and Platelets ≥ 100,000 /µL
* Eastern Cooperative Oncology Group status (ECOG) ≤2 oR Karnofsky ≥80%
* Signed Informed Consent
* Left ventricular ejection fraction (LVEF) >40%
* Normal liver function enzyme tests
* Preserved renal function

Exclusion Criteria:

* Patients not willing to participate or to sign the informed consent
* Patients who do not meet the inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 3 years
  Time between transplantation and relapse or last follow-up

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Time between transplantation and dead or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eucario Leon Rodriguez, M.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Monica M Rivera Franco, M.D.,MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieto Y, Thall P, Valdez B, Andersson B, Popat U, Anderlini P, Shpall EJ, Bassett R, Alousi A, Hosing C, Kebriaei P, Qazilbash M, Frazier E, Gulbis A, Chancoco C, Bashir Q, Ciurea S, Khouri I, Parmar S, Shah N, Worth L, Rondon G, Champlin R, Jones RB. High-dose infusional gemcitabine combined with busulfan and melphalan with autologous stem-cell transplantation in patients with refractory lymphoid malignancies. Biol Blood Marrow Transplant. 2012 Nov;18(11):1677-86. doi: 10.1016/j.bbmt.2012.05.011. Epub 2012 May 27. PMID 22643322
- [Background] Peters GJ, Ruiz van Haperen VW, Bergman AM, Veerman G, Smitskamp-Wilms E, van Moorsel CJ, Kuiper CM, Braakhuis BJ. Preclinical combination therapy with gemcitabine and mechanisms of resistance. Semin Oncol. 1996 Oct;23(5 Suppl 10):16-24. PMID 8893877
- [Background] Wang E, Gulbis A, Hart JW, Nieto Y. The emerging role of gemcitabine in conditioning regimens for hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2014 Sep;20(9):1382-9. doi: 10.1016/j.bbmt.2014.04.025. Epub 2014 May 9. PMID 24816580
- [Background] Anderlini P, Saliba RM, Ledesma C, Chancoco C, Alousi AM, Shpall EJ, Popat UR, Hosing CM, Khouri IF, Nieto Y, Ciurea S, Younes A, Fanale MA, Acholonu S, Valverde R, Champlin RE. Gemcitabine, fludarabine and melphalan as a reduced-intensity conditioning regimen for allogeneic stem cell transplant in relapsed and refractory Hodgkin lymphoma: preliminary results. Leuk Lymphoma. 2012 Mar;53(3):499-502. doi: 10.3109/10428194.2011.615427. Epub 2011 Oct 24. No abstract available. PMID 21859247
- [Background] Matsuda A, Sasaki T. Antitumor activity of sugar-modified cytosine nucleosides. Cancer Sci. 2004 Feb;95(2):105-11. doi: 10.1111/j.1349-7006.2004.tb03189.x. PMID 14965358
- [Background] Spasokoukotskaja T, Arner ES, Brosjo O, Gunven P, Juliusson G, Liliemark J, Eriksson S. Expression of deoxycytidine kinase and phosphorylation of 2-chlorodeoxyadenosine in human normal and tumour cells and tissues. Eur J Cancer. 1995;31A(2):202-8. doi: 10.1016/0959-8049(94)00435-8. PMID 7718326
- [Background] Braakhuis BJ, Ruiz van Haperen VW, Boven E, Veerman G, Peters GJ. Schedule-dependent antitumor effect of gemcitabine in in vivo model system. Semin Oncol. 1995 Aug;22(4 Suppl 11):42-6. PMID 7481844
- [Background] Csoka K, Liliemark J, Larsson R, Nygren P. Evaluation of the cytotoxic activity of gemcitabine in primary cultures of tumor cells from patients with hematologic or solid tumors. Semin Oncol. 1995 Aug;22(4 Suppl 11):47-53. PMID 7481845
- [Background] Plunkett W, Huang P, Searcy CE, Gandhi V. Gemcitabine: preclinical pharmacology and mechanisms of action. Semin Oncol. 1996 Oct;23(5 Suppl 10):3-15. PMID 8893876